CLINICAL TRIAL: NCT00371566
Title: A Randomized, Single Blinded, Placebo-controlled, Multi-centre, Phase II Study of Lapatinib in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: A Study Of Lapatinib Versus Placebo Followed By Chemoradiation In Patients With Locally Advanced Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGF104334
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-04

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: squamous cell carcinoma of head and neck; lapatinib; ErbB1/ErbB2 inhibitor; apoptosis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Lapatinib; Platinum Compounds; Radiotherapy

ARMS (2):
- Lapatinib (Experimental)
  Interventions: Drug: Lapatinib oral tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lapatinib oral tablets
  Other Names: platinum - based chemotherapy; radiotherapy
  Arms: Lapatinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a study comparing the activity of lapatinib versus placebo followed by chemoradiation. This study is designed to explore the effects of lapatinib monotherapy on apoptosis/necrosis, in pre-treatment and post-treatment tumour tissue samples in subjects with locally advanced squamous cell carcinoma of head and neck.

ELIGIBILITY:
Inclusion criteria:

* Willing and able to sign a written informed consent.
* Histologically or cytologically confirmed diagnosis of SCCHN.
* Stage III, IVA and IVB disease will be eligible, who are to receive chemoradiation therapy as primary treatment (total dose ≥ 65 Gy). Subjects with distant metastases (stage IVC) will be excluded.
* Willing and able to have a tumour biopsy taken at screening and a second tumour biopsy taken during lapatinib/placebo administration.
* Male or female ≥18 years of age.

Criteria for female subjects or female partners of male subjects: Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are postmenopausal); Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhoea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at screening and agree to one of the following:

Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or

Consistent and correct use of one of the following acceptable methods of birth control:

male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; implants of levonorgestrel; injectable progestogen; any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progestogen only); or barrier methods, including diaphragm or condom with a spermicide.

* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
* Subjects must have adequate haematological, renal and hepatic function. Calculated creatinine clearance ≥50 ml/min as determined by the method of Cockcroft and Gault [Cockcroft, 1976] or by the EDTA method.

Absolute neutrophil count ≥1,500/μl, platelets ≥100,000/μl. Haemoglobin ≥9gm/dL (5mmol/L). Aspartate (AST) and alanine transaminase (ALT) less than three times the upper limit of the normal range (ULN).

Total bilirubin ≤2.0 mg/dL.

* Left ventricular ejection fraction (LVEF) within the institutional normal ranges as measured by echocardiogram (ECHO) or Multigated Acquisition (MUGA) scans.
* Able to swallow tablet whole or swallow a suspension of the tablet dissolved in water at study inclusion. If necessary, the suspension may be administered via percutaneous endoscopic gastrostomy (PEG), percutaneous jejunostomy tube (JTube), or a nasogastric tube (NG or Dobhoff type tube).
* Life expectancy of at least 6 months as judged by the investigator.

Exclusion criteria:

* Subjects with paranasal sinuses, nasopharyngeal and nasal cavity tumours;
* Subjects who have received prior systemic chemotherapy given with curative intent;
* Subjects who received prior radiotherapy;
* Prior or concurrent treatment with tyrosine kinase inhibitors;
* Use of any investigational agent within 30 days or 5 half-lives, whichever is longer, preceding the first dose of lapatinib;
* Concurrent use of CYP3A4 inducers or inhibitors;
* Subjects with known history of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure;
* History of another malignancy within the last 5 years, with the exception of completely resected basal or squamous cell skin cancer, or successfully treated in situ carcinoma. History of non-invasive lesion or in-situ carcinoma of head and neck that was successfully treated with surgery, photodynamics or laser, will be permitted;
* Distant metastases, ie Stage IVC;
* Females or males of child-bearing potential who are sexually active, if they do not agree to practice an effective method of contraception. (For example oral contraceptives, IUD or diaphragm plus spermicide);
* Pregnant or lactating females (female patients of childbearing potential will undertake pregnancy testing at screening and during study completion/withdrawal visits);
* Malabsorption syndrome, disease significantly affecting GI function, that could affect absorption of lapatinib;
* History of allergic reactions to appropriate diuretics or antiemetics (e.g. 5-HT3 antagonists) to be administered with platinum-based chemotherapy;
* The investigator considers the patient unfit for the study as a result of the medical interview, physical examinations, or screening investigations;
* Subjects taking any prohibited medication (See Section 8.2)

Other Eligibility Criteria Considerations:

To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the following document(s) for detailed information regarding warnings,precautions, contraindications, adverse events, and other significant data pertaining to the investigational product(s) being used in this study: investigator's brochure IB and any IB supplements, and expedited investigator safety reports

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, PhD, Study Director — GlaxoSmithKline
Locations (9):
- France (3):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Athens, Greece
- India (2):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Thiruvananthapuram
- GSK Investigational Site, Lima, Lima Province, Peru
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects who were given Placebo for 2 to 6 weeks followed by 4 weeks of standard treatment of radiotherapy (of more than or equal to 65 Gy) and concurrent platinum-based Chemotherapy (based on the institutions standard of care)
- Lapatinib: Subjects who were given once daily dose of oral lapatinib 1500 mg for 2 -6 weeks, followed by 4 weeks of standard treatment of radiotherapy (of more than or equal to 65 Gy) and concurrent platinum-based chemotherapy (based on the institutions standard care).
Period: Treatment Phase
Arm/Group | Placebo | Lapatinib
Started | 36 | 71
Completed | 36 | 68 (1 screen failure included in the ITT population)
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Chemoradiation Phase
Arm/Group | Placebo | Lapatinib
Started | 36 | 68
Completed | 31 | 65
Not Completed | 5 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non compliant | 0 | 1
Not completed — Progressive Disease | 1 | 1
Not completed — Death | 2 | 0
Period: Follow Up Phase
Arm/Group | Placebo | Lapatinib
Started | 31 | 65
Completed | 28 | 58
Not Completed | 3 | 7
Not completed — Death | 0 | 5
Not completed — Disease progression | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Subjects who were given Placebo for 2 to 6 weeks followed by 4 weeks of standard treatment of radiotherapy (of more than or equal to 65 Gy) and concurrent platinum-based Chemotherapy (based on the intitutions standard of care)
- Total: Total of all reporting groups
Arm/Group | Placebo | Lapatinib | Total
Number analyzed (Participants) | 36 | 71 | 107
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.47) | 57.7 (11.01) | 57.1 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 16 | 20
  Male | 32 | 55 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 39 | 60
  African American | 0 | 0 | 0
  American Indian or Alaska Native | 3 | 11 | 14
  Asian-Central and South Asian Heritage | 9 | 19 | 28
  Asian-Japanese East/South east Heritage | 2 | 2 | 4
  Asian-Mixed Heritage | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Apoptotic Index During Treatment Phase
Description: Apoptotic Index-TUNEL Assay is a method which counts a total of at least 1000 neoplastic nuclei(Cells with morphological changes defining cell death) subdivided in 10 fields chosen randomly at 400x magnification. A 'responder' was defined as having 20% cell death.
Time Frame: Baseline and Week 2
Population: The Intent-to-treat (ITT) population comprised of all subjects who were randomised to study treatment, regardless of whether they actually received study medication.
Measure: Mean (Standard Deviation); unit: Percentage of positive cells
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 27 | 57
Percentage of positive cells | 6.2 (12.10) | 4.2 (5.53)
Statistical Analysis 1: Comparison: Placebo vs Lapatinib; The study was designed to provide evidence to support the null hypothesis: Delta equals 0% or reject it in favor of the two sided alternative hypothesis: Delta does not equal 0%, where Delta was the difference in the true response rate for the two treatment groups; Test type: Superiority or Other; p = .394, ANCOVA; Null hypothesis or reject it in favor of the two sided alternative hypothesis; Mean Difference (Net) = -1.7, 95% CI [-5.50 to 2.19], Standard Deviation 1.93

2. Secondary Outcome: Change From Baseline of Cell Proliferation Rate of the Ki-67 Proliferative Index in Tumour Biopsy Samples During Treatment Phase
Description: The Ki-67 protein is expressed in all phases of the cell cycle except G0 (low level phase) and serves as a good marker for cell proliferation. Scoring is assessed by point counting 500 to 1000 cells, and is reported as percent positive cells. 20% positive cells to define "positive" (i.e. high risk)
Time Frame: Baseline and Week 2
Population: The mITT (modified Intent-to-Treat) population consisted of all subjects who were randomised to study treatment, did not miss lapatinib/placebo treatment for more than 7 consecutive days and had provided sufficient tumor biopsy sample for the primary endpoint analysis.
Measure: Mean (Standard Deviation); unit: Percent of positive cells
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 27 | 57
Percent of positive cells | -1.2 (7.90) | -5.6 (12.53)

3. Secondary Outcome: Overall Radiological Response After Treatment Phase in mITT Population
Description: Over all: Complete Response (CR)- absence of lesions. Partial Response (PR)- CR or PR of target lesions and incomplete response (IC) or stable disease (SD) in other lesions with no new lesions or progressive disease (PD). Stable Disease (SD)-no PD or Response. Progressive Disease (PD)-PD or new lesions. Not Evaluable(NE)- no other definitions. Number of subjects included those who had a scan immediately post lapatanib/placebo monotherapy.
Time Frame: Baseline and End of Treatment (Week 2 - 6)
Population: The mITT population consisted of all subjects who were randomised to study treatment, did not miss lapatinib/placebo treatment for more than 7 consecutive days and had provided sufficient tumour biopsy sample for the primary endpoint analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 12 | 20
Participants
  Complete Response | 0 | 1
  Partial Response | 0 | 3
  Stable Disease | 10 | 12
  Progressive Disease | 2 | 0
  Non-Evaluable | 0 | 4

4. Secondary Outcome: Overall Radiological Response After Follow-up Phase in mITT Population
Description: Over all: Complete Response(CR)-absence of lesions. Partial Response(PR)- CR or PR of target lesions and incomplete response (IC) or stable disease (SD)in other lesions with no new lesions or progressive disease (PD). Stable Disease(SD)-no PD or Response. Progressive Disease(PD)-PD or new lesions. Not Evaluable(NE)- no other definitions. Number of subjects included those who were considered evaluable if they completed a full course of chemoradiotherapy and were able to provide a baseline and follow-up scan following the completion of chemoradiation.
Time Frame: Baseline and End of Follow-up (Week 19 - 25)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 23 | 47
Participants
  Complete Response | 2 | 11
  Partial Response | 13 | 29
  Stable Disease | 2 | 3
  Progressive Disease | 6 | 4

5. Secondary Outcome: Overall Radiological Response After Treatment Phase in ITT Population
Description: Over all: Complete Response (CR)-absence of lesions. Partial Response (PR)- CR or PR of target lesions and incomplete response (IC) or stable disease (SD) in other lesions with no new lesions or progressive disease (PD). Stable Disease (SD)-no PD or Response. Progressive Disease (PD)-PD or new lesions. Not Evaluable(NE)- no other definitions.
Time Frame: Baseline and End of Treatment (Week 2 - 6)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 16 | 24
Participants
  Complete Response | 0 | 1
  Partial Response | 0 | 3
  Stable Disease | 12 | 15
  Progressive Disease | 4 | 0
  Non-Evaluable | 0 | 5

6. Secondary Outcome: Overall Radiological Response After Follow-up Phase in ITT Population
Description: Over all: Complete Response (CR) - absence of lesions. Partial Response (PR) - CR or PR of target lesions and incomplete response (IC) or stable disease (SD) in other lesions with no new lesions or progressive disease (PD). Stable Disease (SD)- no PD or Response. Progressive Disease (PD)- PD or new lesions. Not Evaluable(NE)- no other definitions.
Time Frame: Baseline and End of Follow-up (week 19 - 25)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 30 | 58
Participants
  Complete Response | 2 | 16
  Partial Response | 17 | 34
  Stable Disease | 2 | 4
  Progressive Disease | 9 | 4

7. Secondary Outcome: Number of Circulating Tumor Cells at Baseline in mITT Population
Description: This measures the participants with Circulating Tumor Cells (CTC's)Pre-Treatment numbers of 0 to >= 4. CTC's are tumor cells that escape from the primary tumor into the bloodstream and travel through the circulation to distant sites where they develop into secondary tumors.
Time Frame: Baseline
Population: The mITT population consisted of all subjects who were randomised to study treatment, did not miss lapatinib/placebo treatment for more than 7 consecutive days and had provided sufficient tumour biopsy sample for the primary endpoint analysis. mITT FOLLOW-UP Population of Circulation Tumor Cells
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 12 | 22
Participants
  Number of CTC's 0 | 7 | 18
  Number of CTC's 1 | 2 | 1
  Number of CTC's 2 | 1 | 0
  Number of CTC's 3 | 0 | 0
  Number of CTC's ≥4 | 0 | 1
  No result | 2 | 2

8. Secondary Outcome: Number of Participants With Circulating Tumor Cells After Treatment Phase in mITT Population
Description: This measures the participants with Circulating Tumor Cells (CTC's) after treatment numbers of 0 to >= 4. CTC's are tumor cells that escape from the primary tumor into the bloodstream and travel through the circulation to distant sites where they develop into secondary tumors.
Time Frame: End of Treatment (week 2 - 6)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 13 | 19
Participants
  Number of CTC's 0 | 12 | 13
  Number of CTC's 1 | 0 | 3
  Number of CTC's 2 | 0 | 1
  Number of CTC's 3 | 0 | 0
  Number of CTC's >=4 | 0 | 2
  No result | 1 | 0

9. Secondary Outcome: Number of Participants With Circulating Tumor Cells After Chemoradiotherapy Phase in mITT Population
Description: This measures the participants with Circulating Tumor Cells (CTC's) after chemoradiotherapy numbers of 0 to >= 4. CTC's are tumor cells that escape from the primary tumor into the bloodstream and travel through the circulation to distant sites where they develop into secondary tumors.
Time Frame: End of Chemoradiotherapy (week 10 - 13)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 5 | 2
Participants
  Number of CTC's 0 | 4 | 2
  Number of CTC's 1 | 0 | 0
  Number of CTC's 2 | 0 | 0
  Number of CTC's 3 | 1 | 0
  Number of CTC's >=4 | 0 | 0
  No result | 0 | 0

10. Secondary Outcome: Number of Biomarkers Including ErbB1, ErbB2, pErbB1, and pErb2 at Baseline and During Treatment Phase
Description: Estrogen Receptor (ER) variants, ERB-B2 and ERB B-5 consist of the major proportion of ER expression both in normal and cancer tissues. The exact role of these markers are unknown. Acronyms defined: ICH (immunohistochemical) and FISH (fluorescence in situ hybridization).
Time Frame: Baseline and Week 2
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 27 | 57
Participants
  ErbB1 by IHC-Baseline 0 expressed | 2 | 0
  ErbB1 by IHC-Treatment 0 expressed | 2 | 0
  ErbB1 by IHC-Baseline 1+ expressed | 2 | 2
  ErbB1 by IHC-Treatment 1+ expressed | 1 | 4
  ErbB1 by IHC-Baseline 2+ expressed | 0 | 10
  ErbB1 by IHC-Treatment 2+ expressed | 1 | 5
  ErbB1 by IHC-Baseline 3+ expressed | 23 | 45
  ErbB1 by IHC-Treatment 3+ expressed | 23 | 48
  ErbB1 by FISH-Baseline Amplified | 8 | 17
  ErbB1 by FISH-Treatment Amplified | 0 | 0
  ErbB1 by FISH-Baseline Non Amplified | 19 | 40
  ErbB1 by FISH-Treatment Non Amplified | 0 | 0
  ErbB2 by IHC-Baseline 0 expressed | 19 | 42
  ErbB2 by IHC-Treatment 0 expressed | 15 | 26
  ErbB2 by IHC-Baseline 1+ expressed | 6 | 13
  ErbB2 by IHC-Treatment 1+ expressed | 11 | 29
  ErbB2 by IHC-Baseline 2+ expressed | 2 | 1
  ErbB2 by IHC-Treatment 2+ expressed | 1 | 1
  ErbB2 by IHC-Baseline 3+ expressed | 0 | 1
  ErbB2 by IHC-Treatment 3+ expressed | 0 | 1
  ErbB2 by FISH-Baseline Amplified | 2 | 1
  ErbB2 by FISH-Treatment Amplified | 0 | 0
  ErbB2 by FISH-Baseline Non Amplified | 25 | 54
  ErbB2 by FISH-Treatment Non Amplified | 0 | 2
  pErbB1 by IHC-Baseline 0 expressed | 0 | 3
  pErbB1 by IHC-Baseline 1+ expressed | 13 | 31
  pErbB1 by IHC-Treatment 1+ expressed | 14 | 38
  pErbB1 by IHC-Baseline 2+ expressed | 11 | 18
  pErbB1 by IHC-Treatment 2+ expressed | 11 | 15
  pErbB1 by IHC-Baseline 3+ expressed | 3 | 5
  pErbB1 by IHC-Treatment 3+ expressed | 2 | 1
  pErbB2 by IHC-Baseline 0 expressed | 13 | 25
  pErbB2 by IHC-Treatment 0 expressed | 13 | 24
  pErbB2 by IHC-Baseline 1+ expressed | 12 | 30
  pErbB2 by IHC-Treatment 1+ expressed | 12 | 29
  pErbB2 by IHC-Baseline 2+ expressed | 1 | 1
  pErbB2 by IHC-Treatment 2+ expressed | 1 | 4
  pErbB2 by IHC-Baseline 3+ expressed | 0 | 0
  pErbB2 by IHC-Treatment 3+ expressed | 0 | 0
  pErbB2 by IHC-Baseline - Missing expression | 1 | 1
  pErbB2 by IHC-Treatment Missing expression | 1 | 0

11. Secondary Outcome: Number of Biomarkers Including Tumor Protein 53 and HPV During Treatment Phase
Description: Tumor Suppressor p53 is welcomed and described as "the guardian angel gene," it conserves stability by preventing genome mutation. Human Papillomavirus (HPV) biomarker is un-welcomed and is found to be an important precursor cancers of the head and neck. HPV biomarkers have the ability to bind to and inactivate the Tumor Suppressor p53 biomarker.
Time Frame: Week 2
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 71
Participants
  Tumor Protein 53 - 0 expression | 14 | 25
  Tumor Protein 53 - 1+ expression | 5 | 14
  Tumor Protein 53 - 2+ expression | 3 | 11
  Tumor Protein 53 - 3+ expression | 14 | 19
  Tumor Protein 53 - missing expression | 0 | 0
  HPV - Negative | 36 | 64
  HPV - Positive | 0 | 5

12. Secondary Outcome: Summary of Adverse Events by Maximum Toxicity Grade Started During Treatment Phase
Description: Toxicity Grading scale 0=none, 1=transient symptom, 2=mild symptom that does not interfere with activities of daily living (ADL's) 3=mild but interfers with ADL's w/o hospitalization. 4=requires hopitalization 5=Death.
Time Frame: Week 1 through Week 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Rash - Grade 3 | 0 | 1
  Rash - Grade 4 | 0 | 0
  Rash - Grade 5 | 0 | 0
  Acne - Grade 3 | 0 | 1
  Acne - Grade 4 | 0 | 0
  Acne - Grade 5 | 0 | 0
  Diarrhea - Grade 3 | 0 | 1
  Diarrhea - Grade 4 | 0 | 0
  Diarrhea - Grade 5 | 0 | 0
  Anaemia - Grade 3 | 0 | 1
  Anaemia - Grade 4 | 0 | 0
  Anaemia - Grade 5 | 0 | 0
  Hyperglycaemia - Grade 3 | 1 | 0
  Hyperglycaemia - Grade 4 | 0 | 0
  Hyperglycaemia - Grade 5 | 0 | 0
  Pain in jaw - Grade 3 | 1 | 0
  Pain in jaw - Grade 4 | 0 | 0
  Pain in jaw - Grade 5 | 0 | 0
  Tumor Haemorrhage - Grade 3 | 1 | 0
  Tumor Haemorrhage - Grade 4 | 0 | 0
  Tumor Haemorrhage - Grade 5 | 0 | 0

13. Secondary Outcome: Summary of Adverse Events by Maximum Toxicity Grade (Grade 3 or Higher) Started During or After the Chemoradiotherapy Phase
Description: Toxicity Grading scale 0=none, 1= transient symptom, 2=mild symptom that does not interfere with activities of daily living (ADL's) 3=mild but interfers with ADL's w/o hospitalization. 4=requires hopitalization 5=Death.
Time Frame: Week 10 through 25
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Mucosal Inflamation-Grade 3 | 3 | 24
  Mucosal Inflamation-Grade 4 | 0 | 2
  Mucosal Inflamation-Grade 5 | 0 | 0
  Skin Reaction-Grade 3 | 3 | 6
  Skin Reaction-Grade 4 | 0 | 1
  Skin Reaction-Grade 5 | 0 | 0
  Neutropenia-Grade 3 | 3 | 4
  Neutropenia-Grade 4 | 1 | 0
  Neutropenia-Grade 5 | 0 | 0
  Asthenia-Grade 3 | 2 | 3
  Asthenia-Grade 4 | 0 | 0
  Asthenia-Grade 5 | 0 | 0
  Soft Tissue Inflamation-Grade 3 | 1 | 2
  Soft Tissue Inflamation-Grade 4 | 0 | 0
  Soft Tissue Inflamation-Grade 5 | 0 | 0
  Odynophagia-Grade 3 | 2 | 2
  Odynophagia-Grade 4 | 0 | 0
  Odynophagia-Grade 5 | 0 | 0
  General Physical Health deterioration-Grade 3 | 0 | 2
  General Physical Health deterioration-Grade 4 | 0 | 0
  General Physical Health deterioration-Grade 5 | 0 | 0
  Rash-Grade 3 | 0 | 2
  Rash-Grade 4 | 0 | 0
  Rash-Grade 5 | 0 | 0
  Radiation Skin Injury-Grade 3 | 0 | 2
  Radiation Skin Injury-Grade 4 | 0 | 0
  Radiation Skin Injury-Grade 5 | 0 | 0
  Dysphagia-Grade 3 | 3 | 1
  Dysphagia-Grade 4 | 0 | 0
  Dysphagia-Grade 5 | 0 | 0
  Nausea-Grade 3 | 1 | 1
  Nausea-Grade 4 | 0 | 0
  Nausea-Grade 5 | 0 | 0
  Stomatitis-Grade 3 | 1 | 1
  Stomatitis-Grade 4 | 0 | 0
  Stomatitis-Grade 5 | 0 | 0
  Radiation mucositis-Grade 3 | 2 | 1
  Radiation mucositis-Grade 4 | 0 | 0
  Radiation mucositis-Grade 5 | 0 | 0
  Weight decrease-Grade 3 | 1 | 1
  Weight decrease-Grade 4 | 0 | 0
  Weight decrease-Grade 5 | 0 | 0
  Pain-Grade 3 | 0 | 1
  Pain-Grade 4 | 0 | 0
  Pain-Grade 5 | 0 | 0
  Constipation-Grade 3 | 0 | 1
  Constipation-Grade 4 | 0 | 0
  Constipation-Grade 5 | 0 | 0
  Skin Ulcer-Grade 3 | 0 | 1
  Skin Ulcer-Grade 4 | 0 | 0
  Skin Ulcer-Grade 5 | 0 | 0
  Dysphonia-Grade 3 | 0 | 1
  Dysphonia-Grade 4 | 0 | 0
  Dysphonia-Grade 5 | 0 | 0
  Leucopenia-Grade 3 | 2 | 1
  Leucopenia-Grade 4 | 0 | 0
  Leucopenia-Grade 5 | 0 | 0
  AST increase-Grade 3 | 0 | 1
  AST increase-Grade 4 | 0 | 0
  AST increase-Grade 5 | 0 | 0
  Trimus-Grade 3 | 0 | 1
  Trimus-Grade 4 | 0 | 0
  Trimus-Grade 5 | 0 | 0
  Bipolar disorder-Grade 3 | 0 | 1
  Bipolar disorder-Grade 4 | 0 | 0
  Bipolar disorder-Grade 5 | 0 | 0
  Diplopia-Grade 3 | 0 | 1
  Diplopia-Grade 4 | 0 | 0
  Diplopia-Grade 5 | 0 | 0
  Peripheral Embolism-Grade 3 | 0 | 1
  Peripheral Embolism-Grade 4 | 0 | 0
  Peripheral Embolism-Grade 5 | 0 | 0
  Renal Failure-Grade 3 | 0 | 1
  Renal Failure-Grade 4 | 0 | 0
  Renal Failure-Grade 5 | 0 | 0
  Localized edema-Grade 3 | 1 | 0
  Localized edema-Grade 4 | 0 | 0
  Localized edema-Grade 5 | 0 | 0
  Vomiting-Grade 3 | 3 | 0
  Vomiting-Grade 4 | 0 | 0
  Vomiting-Grade 5 | 0 | 0
  Respiratory failure-Grade 3 | 1 | 0
  Respiratory failure-Grade 4 | 0 | 0
  Respiratory failure-Grade 5 | 0 | 0
  Respiratory tract infection-Grade 3 | 1 | 0
  Respiratory tract infection-Grade 4 | 0 | 0
  Respiratory tract infection-Grade 5 | 0 | 0
  Sepsis-Grade 3 | 1 | 0
  Sepsis-Grade 4 | 0 | 0
  Sepsis-Grade 5 | 0 | 0
  Staphyloccocal sepsis-Grade 3 | 0 | 0
  Staphyloccocal sepsis-Grade 4 | 0 | 0
  Staphyloccocal sepsis-Grade 5 | 1 | 0
  Hyponatraemia-Grade 3 | 2 | 0
  Hyponatraemia-Grade 4 | 0 | 0
  Hyponatraemia-Grade 5 | 0 | 0
  Hypernatraemia-Grade 3 | 0 | 0
  Hypernatraemia-Grade 4 | 0 | 1
  Hypernatraemia-Grade 5 | 0 | 0
  Ketoacidosis-Grade 3 | 1 | 0
  Ketoacidosis-Grade 4 | 0 | 0
  Ketoacidosis-Grade 5 | 0 | 0
  Post Procedural Haemorrhage-Grade 3 | 1 | 0
  Post Procedural Haemorrhage-Grade 4 | 0 | 0
  Post Procedural Haemorrhage-Grade 5 | 0 | 0
  Blood Creatinine Increased-Grade 3 | 1 | 0
  Blood Creatinine Increased-Grade 4 | 0 | 0
  Blood Creatinine Increased-Grade 5 | 0 | 0
  Haematocrit decreased-Grade 3 | 1 | 0
  Haematocrit decreased-Grade 4 | 0 | 0
  Haematocrit decreased-Grade 5 | 0 | 0
  Haemoglobin decreased-Grade 3 | 1 | 0
  Haemoglobin decreased-Grade 4 | 0 | 0
  Haemoglobin decreased-Grade 5 | 0 | 0
  Back Pain-Grade 3 | 1 | 0
  Back Pain-Grade 4 | 0 | 0
  Back Pain-Grade 5 | 0 | 0
  Deep Vein Thrombosis-Grade 3 | 1 | 0
  Deep Vein Thrombosis-Grade 4 | 0 | 0
  Deep Vein Thrombosis-Grade 5 | 0 | 0
  Ventricular Fibrillation-Grade 3 | 0 | 0
  Ventricular Fibrillation-Grade 4 | 0 | 0
  Ventricular Fibrillation-Grade 5 | 1 | 0
  Intestinal Perforation-Grade 3 | 0 | 0
  Intestinal Perforation-Grade 4 | 0 | 0
  Intestinal Perforation-Grade 5 | 0 | 1
  Dyspnoea-Grade 3 | 0 | 0
  Dyspnoea-Grade 4 | 0 | 1
  Dyspnoea-Grade 5 | 0 | 0
  Anaemia-Grade 3 | 0 | 0
  Anaemia-Grade 4 | 0 | 2
  Anaemia-Grade 5 | 0 | 0
  Lymphopenia-Grade 3 | 1 | 0
  Lymphopenia-Grade 4 | 0 | 0
  Lymphopenia-Grade 5 | 0 | 0
  Cardio-respiratory arrest-Grade 3 | 0 | 0
  Cardio-respiratory arrest-Grade 4 | 0 | 0
  Cardio-respiratory arrest-Grade 5 | 0 | 1
  Sudden Death-Grade 3 | 0 | 0
  Sudden Death-Grade 4 | 0 | 0
  Sudden Death-Grade 5 | 0 | 1
  Dry Mouth-Grade 3 | 1 | 0
  Dry Mouth-Grade 4 | 0 | 0
  Dry Mouth-Grade 5 | 0 | 0

14. Secondary Outcome: Comparison of Overall Response During Treatment Phase Using CT/MRI and PET Information
Description: Position Emission Tomography (PET) scans 3-D images are read alongside CT or magnetic resonance imaging (MRI) scans, the combination gives both anatomic and metabolic information. CT = Computerized axial tomography; a type of x-ray for dense areas of the body. MRI = Magnetic Resonance Imaging which captures a picture using Magnets. Better = improvement in response, Worse = response was downgraded.
Time Frame: Week 2 - 4
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 11 | 14
Participants
  Better | 2 | 3
  Same | 8 | 6
  Worse | 0 | 3
  Any Unknown | 0 | 0
  Missing | 1 | 0
  Not Evaluable | 0 | 2

15. Secondary Outcome: Comparison of Overall Response During Follow up Phase Using CT/MRI and PET Information
Description: as for outcome 14
Time Frame: weeks 19 - 25
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 13 | 17
Participants
  Better | 0 | 2
  Same | 11 | 10
  Worse | 1 | 5
  Any Unknown | 0 | 0
  Missing | 1 | 0
  Not Evaluable | 0 | 0

16. Secondary Outcome: Summary of Adverse Events Experienced by 15% or More Subjects in Either Treatment Group
Description: Definition of an adverse event is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Week 1 through 25
Population: Safety population consisted of all randomized subjects who took at least one dose of study medication. This population was based on the actual treatment received, if different to the randomized treatment allocation.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Mucosal Inflammation | 24 | 48
  Odynophagia | 13 | 23
  Asthenia | 17 | 21
  Dysphagia | 12 | 21
  Nausea | 8 | 20
  Vomiting | 13 | 17
  Dry Mouth | 8 | 15
  Neutropenia | 10 | 13
  Radiation Skin Injury | 8 | 13
  Constipation | 8 | 12
  Skin Reaction | 7 | 11
  Pharyngolaryngeal Pain | 6 | 11
  Anorexia | 11 | 10
  Dysphonia | 8 | 8
  Pyrexia | 6 | 6
  Leukopenia | 7 | 3

17. Secondary Outcome: Summary of Fatal/Serious Adverse Events During or After Chemoradiotherapy Phase
Description: Events which started during or After the Chemoradiotherapy Phase. Definition of a serious adverse event is any untoward medicinal occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other.
Time Frame: Week 10 through 25
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Cardio-respiratory arrest | 0 | 1
  Intestinal perforation | 0 | 1
  Respiratory tract infection | 0 | 1
  Sudden death | 0 | 1
  Ventricular fibrillation | 1 | 0

18. Secondary Outcome: Summary of Serious Adverse Events During or After Chemoradiotherapy Phase
Description: Events which started during or After Chemoradiotherapy Phase. Definition of a serious adverse event is any untoward medicinal occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other.
Time Frame: Week 10 through 25
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Mucosal inflammation | 2 | 3
  Constipation | 0 | 2
  Asthenia | 0 | 1
  Bipolar disorder | 0 | 1
  Cardio-respiratory arrest | 0 | 1
  Chronic obstructive pulmonary disease | 0 | 1
  Dehydration | 0 | 1
  General physical health deterioration | 0 | 1
  Intestinal perforation | 0 | 1
  Peripheral embolism | 0 | 1
  Renal failure | 0 | 1
  Respiratory tract infection | 2 | 1
  Skin ulcer | 0 | 1
  Sudden death | 0 | 1
  Electrolyte imbalance | 1 | 0
  Diabetic ketoacidosis | 1 | 0
  Ketoacidosis | 1 | 0
  Lobar pneumonia | 1 | 0
  Neutropenia | 1 | 0
  Parotitis | 1 | 0
  Pneumonia aspiration | 1 | 0
  Post procedural haemorrhage | 1 | 0
  Pyrexia | 2 | 0
  Renal Impairment | 1 | 0
  Sepsis | 1 | 0
  Septic shock | 1 | 0
  Upper respiratory tract infection | 1 | 0
  Ventricular fibrillation | 1 | 0
  Vomiting | 2 | 0
  Weight decreased | 1 | 0

19. Secondary Outcome: Adverse Events by Maximum Toxicity Grade 3 During or After Chemoradiotherapy Phase
Description: Events which started during or after Chemoradiotherapy Phase. "Grade 3" are severe and undesirable Adverse Event (significant symptoms requiring hospitalization or invasive intervention; transfusion; elective interventional radiological procedure; therapeutic endoscopy or operation).
Time Frame: Week 10 through 25
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Mucosal inflammation | 9 | 24
  Skin reaction | 3 | 6
  Neutropenia | 3 | 4
  Asthenia | 2 | 3
  Soft tissue inflammation | 1 | 2
  Odynophagia | 2 | 2
  General physical health deterioration | 0 | 2
  Rash | 0 | 2
  Radiation skin injury | 0 | 2
  Dysphagia | 3 | 1
  Nausea | 1 | 1
  Stomatitis | 1 | 1
  Radiation mucositis | 2 | 1
  Weight decreased | 1 | 1
  Pain | 0 | 1
  Constipation | 0 | 1
  Skin ulcer | 0 | 1
  Dysphonia | 0 | 1
  Leucopenia | 2 | 1
  Aspartate aminotransferase increased | 0 | 1
  Trismus | 0 | 1
  Bipolar disorder | 0 | 1
  Diplopia | 0 | 1
  Peripheral embolism | 0 | 1
  Renal failure | 0 | 1
  Localised oedema | 1 | 0
  Vomiting | 3 | 0
  Respiratory failure | 1 | 0
  Respiratory tract infection | 1 | 0
  Sepsis | 1 | 0
  Hyponatraemia | 2 | 0
  Ketoacidosis | 1 | 0
  Post procedural haemorrhage | 1 | 0
  Blood creatinine increased | 1 | 0
  Haematocrit decreased | 1 | 0
  Haemoglobin decreased | 1 | 0
  Back pain | 1 | 0
  Deep vein thrombosis | 1 | 0
  Lymphopenia | 1 | 0
  Dry mouth | 1 | 0

20. Secondary Outcome: Adverse Events (AEs) by Maximum Toxicity Grade 4 During or After Chemoradiotherapy Phase
Description: Events which started during or after Chemoradiotherapy Phase. "Grade 4" are life-threatening or disabling Adverse Event (complicated by acute, life-threatening metabolic or cardiovascular complications such as circulatory failure, hemorrhage, sepsis. Life-threatening physiologic consequences; need for intensive care or emergent invasive procedure; emergent interventional radiological procedure, therapeutic endoscopy or operation).
Time Frame: Week 10 through 25
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Mucosal inflammation | 0 | 2
  Skin reaction | 0 | 1
  Neutropenia | 1 | 0
  Hypernatraemia | 0 | 1
  Dyspnoea | 0 | 1
  Anaemia | 0 | 2

21. Secondary Outcome: Adverse Events by Maximum Toxicity Grade 5 During or After Chemoradiotherapy Phase
Description: Events which started during or after Chemoradiotherapy Phase. "Grade 5" are death related to Adverse Event.
Time Frame: Week 10 through 25
Population: as for outcome 16
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 36 | 69
Participants
  Respiratory tract infection | 0 | 1
  Staphyloccocal sepsis | 1 | 0
  Ventricular fibrillation | 1 | 0
  Intestinal perforation | 0 | 1
  Cardio-respiratory arrest | 0 | 1
  Sudden death | 0 | 1

22. Secondary Outcome: Relative Change From Baseline of Ktrans Median (1/Min) After 2 - 4 Weeks of Treatment
Description: Dynamic Contrast enhanced Magnetic Resonance Imaging (DCE-MRI) tracks the diffusion of an administered contrast agent from -intra into the extravascular tissue over time. Ktrans estimates blood flow and relates to the ease of exchange into extravascular spaces. A volume transfer (i.e, 1/min) constant of contrast agent is used to determine vascular permeability. By plugging DCE-MRI results into an appropriate pharmacokinetic model, physiological parameters of the tumor (e.g.,tissue perfusion, vessel permeability, vascular surface area, and extracellular/vascular volume fraction) are determined.
Time Frame: Baseline, and Week 2 - 4
Population: The mITT population consisted of all subjects who were randomised to study treatment, did not miss lapatinib/placebo treatment for more than 7 consecutive days and had provided sufficient tumour biopsy sample for the primary endpoint analysis. DCE-MRI population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -2.70 (25.364) | 6.15 (22.792)

23. Secondary Outcome: Relative Change From Baseline of Kep Mean (1/Min) After 2 - 4 Weeks of Treatment
Description: DCE-MRI tracks the diffusion of an intravascularly administered contrast agent into the extravascular tissue over time. Over a period of time, the contrast agent diffuses back into the vasculature (described by the rate constant or Kep). The lower the Kep, the longer the contrast remains in the extravascular space and is more prolonged. A volume transfer (i.e, 1/min) constant of contrast agent is used to determine vascular permeability. By plugging DCE-MRI results into an appropriate pharmacokinetic model, physiological parameters of the tumor (e.g., vessel permeability, etc.) are determined.
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | 10.30 (33.630) | -14.54 (8.898)

24. Secondary Outcome: Relative Change From Baseline of Kep Perfused (1/Min) After 2 - 4 Weeks of Treatment
Description: as for outcome 23
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | 7.63 (26.965) | -19.96 (8.662)

25. Secondary Outcome: Relative Change From Baseline of Kep Whole (1/Min) After 2 - 4 Weeks of Treatment
Description: as for outcome 23
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | 8.87 (29.875) | -19.64 (6.716)

26. Secondary Outcome: Relative Change From Baseline of Ktrans Mean (1/Min) After 2 - 4 Weeks of Treatment
Description: as for outcome 22
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -1.90 (27.965) | 4.02 (17.683)

27. Secondary Outcome: Relative Change From Baseline of Ktrans Perfused (1/Min) After 2 - 4 Weeks of Treatment
Description: as for outcome 22
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -1.44 (23.029) | 0.69 (34.213)

28. Secondary Outcome: Relative Change From Baseline of Ktrans Whole (1/Min) After 2 - 4 Weeks of Treatment
Description: as for outcome 22
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -2.02 (20.971) | 0.30 (31.783)

29. Secondary Outcome: Relative Change From Baseline of IAUC Median (90) After 2 - 4 Weeks of Treatment
Description: Dynamic Contrast - enhanced Magnetic Resonance Imaging (DCE-MRI) tracks the diffusion of an intravascularly administered contrast agent from intravascular into the extravascular tissue over time. Initial area under the contrast (IAUC), tracks the concentration versus time curve 90 seconds after contrast injection (IAUC90). By plugging DCE-MRI results into an appropriate pharmacokinetic model, physiological parameters of the tumor microenvironment (e.g., tissue perfusion, vessel permeability, vascular surface area, and extracellular-extra vascular volume fraction) are determined.
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -2.07 (30.188) | 14.08 (23.998)

30. Secondary Outcome: Relative Change From Baseline of IAUC Mean (90) After 2 - 4 Weeks of Treatment
Description: as for outcome 29
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -3.30 (28.415) | 13.48 (20.763)

31. Secondary Outcome: Relative Change From Baseline of Perfused IAUC (90) After 2 - 4 Weeks of Treatment
Description: as for outcome 29
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -2.40 (29.521) | 12.57 (28.722)

32. Secondary Outcome: Relative Change From Baseline of Whole IAUC(90) After 2 - 4 Weeks of Treatment
Description: as for outcome 29
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | -2.43 (29.313) | 12.52 (28.974)

33. Secondary Outcome: Relative Change From Baseline of Kep Median (1/Min) After 2 - 4 Weeks of Treatment
Description: as for outcome 23
Time Frame: Baseline, and Week 2 - 4
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Lapatinib
Number analyzed (Participants) | 6 | 4
Percent change | 2.88 (19.177) | -9.32 (10.002)

ADVERSE EVENTS:
Time Frame: Started prior to and during Lapatanib/Placebo phase, during or after chemoradiotherapy phase.
Description: Safety population used in this analysis consisting of all randomized subjects who took at least one dose of study medication. This population was based on the actual treatment received, if different to the randomized treatment allocation.
Groups:
- Lapatinib: Subjects who were given once daily dose of oral lapatinib 1500 mg for 2 -6 weeks, followed by 4 weeks of standard treatment of radiotherapy (of mor than or equal to 65 Gy) and concurrent platinum-based chemotherapy (based on the institutions standard care).
Arm/Group | Placebo | Lapatinib
Serious Adverse Events (participants affected / at risk) | 14/36 | 14/69
Other Adverse Events (participants affected / at risk) | 36/36 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Lapatinib (N=69)
Pyrexia (Infections and infestations) | 2 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal strangulated hernia (Musculoskeletal and connective tissue disorders) | 1 | 0
Mucosal Inflammation (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthenia (Musculoskeletal and connective tissue disorders) | 0 | 1
General Physical Health deterioration (General disorders) | 0 | 1
Sudden Death (Investigations) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Dehydration (General disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bipolar Disorder (Psychiatric disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral Embolism (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Lobar Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Sepsis (Blood and lymphatic system disorders) | 1 | 0
Septic Shock (Blood and lymphatic system disorders) | 1 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Pneumonia Aspirations (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Weight Decrease (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Lapatinib (N=69)
Mucosal inflammation (Gastrointestinal disorders) | 24 | 48
Asthenia (Musculoskeletal and connective tissue disorders) | 17 | 23
Odynophagia (Gastrointestinal disorders) | 13 | 23
Dysphagia (Gastrointestinal disorders) | 13 | 22
Nausea (Gastrointestinal disorders) | 9 | 21
Rash (Skin and subcutaneous tissue disorders) | 5 | 21
Vomiting (Gastrointestinal disorders) | 14 | 18
Diarrhoea (Gastrointestinal disorders) | 2 | 18
Dry Mouth (Gastrointestinal disorders) | 8 | 15
Anorexia (Metabolism and nutrition disorders) | 11 | 14
Neutropenia (Blood and lymphatic system disorders) | 10 | 13
Radiation Skin Injury (Injury, poisoning and procedural complications) | 8 | 13
Constipation (Gastrointestinal disorders) | 9 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pain (General disorders) | 6 | 8
Pyrexia (General disorders) | 6 | 7
Soft tissue inflammation (General disorders) | 3 | 5
Oedema (General disorders) | 2 | 3
Face oedema (General disorders) | 3 | 1
Oral pain (Gastrointestinal disorders) | 3 | 10
Stomatitis (Gastrointestinal disorders) | 2 | 5
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 3
Aptyalism (Gastrointestinal disorders) | 0 | 5
Toothache (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Mouth hemorrhage (Gastrointestinal disorders) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 7 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Candidiasis (Infections and infestations) | 4 | 4
Oral candidiasis (Infections and infestations) | 2 | 5
Respiratory tract infection (Infections and infestations) | 3 | 1
Oropharyngeal candidiasis (Infections and infestations) | 3 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Anemia (Blood and lymphatic system disorders) | 5 | 10
Leukopenia (Blood and lymphatic system disorders) | 7 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5
Weight decreased (Blood and lymphatic system disorders) | 5 | 9
Blood creatinine increased (Blood and lymphatic system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 4 | 11
Headache (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 4 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 3 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 5
Hypoacusis (Ear and labyrinth disorders) | 2 | 7
Ear pain (Ear and labyrinth disorders) | 4 | 2
Tinnitus (Ear and labyrinth disorders) | 3 | 1
Pallor (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
: GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.